CLINICAL TRIAL: NCT06408090
Title: Knowledge of and Attitudes Toward Hospice, Decision-making Around Hospice in Older Black Adults
Brief Title: Underutilization of Hospice Care in Older Black Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 23-0899
Record Dates: First submitted 2023-10-31; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Hospice Care; Decision Aid; Decision-Making; Aging; Knowledge; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): 200 participants reviewed the PtDA decision tool for education on hospice care and subsequently completed a second survey which was identical to the first.
  Interventions: Other: IDECIDE-HOSPICE
- Interview (Other): 20 of the 200 Intervention participants will complete an interview using qualitative methods surrounding the topic of hospice care and the PtDA.
  Interventions: Other: IDECIDE-HOSPICE
- Control (No Intervention): 200 of the 400 participants completed two identical surveys one month apart but did NOT review the PtDA decision tool prior to completing the second survey timepoint. Instead, these participants reviewed an 8-page attention control activity booklet. These participants are used as a control group in assessing any change in knowledge or opinions of hospice after the intervention group reviewed the PtDA.

INTERVENTIONS:
Other: IDECIDE-HOSPICE — 12-pg educational booklet detailing information about hospice including what hospice is, why someone would use hospice, who pays for hospice, and where hospice services are delivered
  Other Names: PtDA
  Arms: Intervention; Interview

SUMMARY:
This study will sample older Black adults to test their knowledge and opinions of hospice.

DETAILED DESCRIPTION:
Short stays in hospice strain the Medicare system. Black adults over age 65 are one of the fastest growing groups in the US. Despite greater disease burden than their White peers, older Black adults are less likely to enroll in hospice. Misconceptions about hospice and mistrust may contribute to this disparity. The research will seek to understand older Black adults' decision-making processes around hospice. The PtDA is a tool to assist in this decision-making process. The influence of this tool will be measured as well. The sample of older Black adults will represent the national population. The research will explore various subgroups, which previous research has been unable to address. This study will use four validated survey batteries. About 200 of the 400 participants will also review the decision aid. These adults will complete a second survey. About 20 of these adults will also complete an interview about the decision aid. Through the surveys and interviews, this research will explore barriers to hospice usage for older Black adults.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as Black or African American
* Can read and write English

Exclusion Criteria:

* Unable to read/write English
* Have a cognitive impairment that prevents them from providing informed consent

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospice Knowledge | June 2023 through September 2023
  assessed using 23-item hospice knowledge survey
Hospice Beliefs and Attitudes | June 2023 through September 2023
  measured using 8-item Hospice Beliefs and Attitudes Scale (HBAS)
Self-Efficacy | June 2023 through September 2023
  assessed using 11-item Decision Self-Efficacy Scale (DSE)

SECONDARY OUTCOMES:
Medical Mistrust | June 2023 through September 2023
  measured using 17-item Medical Mistrust Index (MMI)

CONTACTS AND LOCATIONS:
Overall Officials: Channing E Tate, PhD, MPH, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT06408090/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT06408090/ICF_001.pdf